CLINICAL TRIAL: NCT06383468
Title: a Randomized Double-blind, Placebo-controlled, Multicenter Phase III Clinical Study to Evaluate the Efficacy and Safety of AK120 in the Treatment of Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Phase III Study to Evaluate the Efficacy and Safety of AK120 in Patients With Moderate to Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK120-301
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK120 600mg/300mg (Experimental): AK120 600mg(first day) then 300mg Q2W subcutaneous injection thereafter until week 50.
  Interventions: Drug: AK120
- Placebo/AK120 600mg to 300mg (Placebo Comparator): placebo Q2W SC, then AK120 600mg at week 16, thereafter change to AK120 300mg Q2W subcutaneous injection until week 50.
  Interventions: Drug: AK120

INTERVENTIONS:
Drug: AK120 — 300mg Q2W subcutaneous injection thereafter until week 50.

SUMMARY:
This is a randomized double-blind, placebo-controlled, multicenter phase III clinical study evaluating the efficacy and safety of AK120 injection in the treatment of patients with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
This is a randomized double-blind, placebo-controlled, multicenter phase III clinical study evaluating the efficacy and safety of AK120 injection in the treatment of patients with moderate to severe atopic dermatitis. The entire study included a screening period, a double-blind controlled treatment period, a conversion and maintenance treatment period, and a safe follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18≤75 years old.
2. Atopic dermatitis (AD) diagnosed at least 1 year before screening.
3. Subject with eczema area and severity index (EASI) score ≥16, Investigator Global Assessment (IGA) score≥ 3, Body Surface Area (BSA) score ≥ 10% at screening and baseline.
4. Previously received at least 4 weeks of moderate to strong or at least 2 weeks of strong local glucocorticoid (TCS) treatment for AD before screening, with poor efficacy or intolerable

Exclusion Criteria:

1. Acute onset of AD within the first 4 weeks of randomization.
2. Have participated in any clinical research on AK120 in the past
3. Received systemic corticosteroids, immunosuppressive/immunomodulatory drugs, phototherapy within the 4 weeks before randomization.
4. Received treatment with other clinical research drugs (non-biological agents) within the first 4 weeks or 5 half-lives of randomization (whichever is longer)
5. Received or planned to receive live vaccine treatment within the 3 months before randomization or during the study period.
6. Received allergen specific immunotherapy within the 3 months before randomization.
7. Have a history of allergies to any component of AK120 and/or severe allergic reactions to monoclonal antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who achieved (Eczema Area and Severity Index) EASI-75 | at week 16
  Percentage of patients in both treatment group and placebo group who achieved EASI 75 at week 16.

SECONDARY OUTCOMES:
Percentage of subjects who achieved 0/1 in the (Investigator's Global Assessment) IGA | at week 16
  The percentage of patients in both treatment group and placebo group who achieved IGA 0/1 score at week 16.

CONTACTS AND LOCATIONS:
Locations (59):
- China (59):
  - Beijing Friendship Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Luhe Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing Three Gorges Medical College Affiliated People's Hospital, Chongqing, Chongqing Municipality
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second Affiliated Hospital of Xiamen Medical College, Xiamen, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Southern Medical University Dermatology Hospital/Guangdong Provincial Dermatology Hospital, Guangzhou, Guangdong
  - Southern Medical University Southern Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Yuebei People's hospital, Guangdong, China, Shaoguan, Guangdong
  - Shunde Hospital of Southern Medical University, Shunde, Guangdong
  - Guangdong Medical University Affiliated Hospital, Zhanjiang, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - Hainan Provincial Fifth People's Hospital, Haikou, Hainan
  - The First Affiliated Hospital of Hainan Medical College, Haikou, Hainan
  - Chengde Medical College Affiliated Hospital, Chengde, Hebei
  - The Second Affiliated Hospital of Xingtai Medical College, Xingtai, Hebei
  - Harbin Medical University Affiliated Second Hospital, Harbin, Heilongjiang
  - Heilongjiang Provincial Hospital, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Renmin Hospital of Wuhan University Hubei General Hospital, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - Changde First People's Hospital, Changde, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of South China University, Hengyang, Hunan
  - Inner Mongolia Medical University Affiliated Hospital, Hohhot, Inner Mongolia
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Jiangsu
  - Changzhou First People's Hospital, Changzhou, Jiangsu
  - Yancheng First People's Hospital, Yancheng, Jiangsu
  - Jiangsu University Affiliated Hospital, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Gannan Medical College, Ganzhou, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Panjin Liaoyou Gemstone Flower Hospital, Panjin, Liaoning
  - Shenyang Integrated Traditional Chinese and Western Medicine Hospital, Shenyang, Liaoning
  - Zhongyi Northeast International Hospital, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Provincial Dermatology Hospital, Jinan, Shandong
  - Shandong University Qilu Hospital, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality
  - Baoji Central Hospital, Baoji, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Institute of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Uygur Autonomous Region People's Hospital, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jiaxing First People's Hospital, Jiaxing, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Ningbo Huamei Hospital, University of Chinese Academy of Sciences, Ningbo, Zhejiang
  - Wenzhou Medical University First Affiliated Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No